CLINICAL TRIAL: NCT03331614
Title: A Randomized Controlled Evaluation of the Effect of Sequential Contraction Compression Device on the Symptomatology of Painful Diabetic Neuropathy (PDN)
Brief Title: An Evaluation of an SCCD on the Symptomatology of Painful DPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rosenblum, Jonathan I., DPM (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCN-1
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Subjects will be sequentially divided into a control group or an active treatment group.
Who Masked: Outcomes Assessor
Masking Description: The data collected by the investigator will be submitted to the assessor without indication of which group is active and which is control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (No Intervention): This group will continue with their current treatment regimen during the course of the study. They will be monitored with daily questionnaires, and at the end of trial visit will also undergo a QST evaluation.
- Active Treatment Group (Active Comparator): This group will continue with their current treatment regimen during the course of the study. In addition they will be given an active intervention with the Flowaid FA-100 SCCD device to utilize at home daily. They will be monitored with daily questionnaires, and at the end of trial visit will also undergo a QST evaluation.
  Interventions: Device: Flowaid FA-100 SCCD

INTERVENTIONS:
Device: Flowaid FA-100 SCCD — The SCCD is a contained external non invasive electric muscle pump. The device attaches to the rear of the calf with 4 electrodes.
  Arms: Active Treatment Group

SUMMARY:
This is a controlled trial to evaluate the efficacy of an Sequential Contraction Compression Device (SCCD) on the symptomatology of Painful Diabetic Neuropathy. Subjects will be divided into a control group where they will be monitored while continuing with their current treatment regimen and into a treatment group where they will continue with their current regimen and have SCCD therapy added. Subjects will be evaluated for Subjective Pain levels, quality of life, breakthrough drug use, sleep levels, and objectively with a Quantitative Sensory Testing device. The trial duration is 30 days.

DETAILED DESCRIPTION:
This is a controlled trial of 30 days duration to evaluate the efficacy of an Sequential Contraction Compression Device (SCCD) on the symptomatology of Painful Diabetic Neuropathy. Subjects will have to have been on a sustained drug regimen for more than 30 days and have an average pain level of 4 on a VAS. Subjects will be divided into a control group where they will be monitored while continuing with their current treatment regimen and into a treatment group where they will continue with their current regimen and have SCCD therapy added. Patients will be asked to use the SCCD device daily on both their legs. Subjects will be evaluated for Subjective Pain levels using a Visual Analog Scale, quality of life using various questionnaires, breakthrough drug use in a daily log, sleep levels i.e. how many consecutive hours of sleep, and objectively with a Quantitative Sensory Testing device.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of Type I or Type II Diabetes Mellitus
* Have a documented diagnosis of Diabetic Peripheral Neuropathy by either their Primary Care Physician or other physician treating their condition made no less than 6 months prior to initiation of the study.
* Have been on stable pain medications (no change to type, dose or frequency) for at least 1 month prior to their entry into the study.Give appropriate written informed consent prior to participation in the study
* Be between 18 and 90 years of age, inclusive, on the day the Informed Consent Form is signed
* Have an average baseline VAS score of 4 or more as assessed during the week just prior to randomization
* Be in reasonable metabolic control, exhibited by HbA1C values of less than 12% as observed by serum test results obtained within 3 months prior to the Screening Visit
* Be willing to remain on the same pain medication regimen for the duration of the study
* If subject is of childbearing potential, she must be using an acceptable method of birth control. Women not of childbearing potential are defined as either surgically sterile or post-menopausal. Post-menopausal women are defined as those women with a documented menstruation cessation for 12 consecutive months prior to signing the Informed Consent Form.
* Subject and caregiver, if applicable, must be accessible and willing to comply with all requirements of the study protocol for the duration of the study.

Exclusion Criteria:

* Clinical evidence of compromised skin (e.g., wound, infection, gangrene) on the lower legs
* Active Charcot's foot on either limb
* Malnourished as evidenced by a pre-albumin of < 11 mg/dL
* Pregnancy or lactating
* Known history of alcohol or drug abuse within the previous one year
* Previous treatment with SCCD
* Elective osseous procedures performed to either foot 30 days prior to Screening visit
* Vascular procedures performed 30 days prior to Screening Visit
* History of poor compliance to medical treatment regimens
* Conditions that may severely compromise their ability to complete the study.
* Concomitant history of Peripheral Arterial disease with an ABI of <0.5
* Chronic pain due to an etiology other than diabetic neuropathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Subjective Pain | 30 days
  Reduction in pain as measured using a pain descriptive Visual Analog Scale (VAS). The SCCD treatment will be considered effective if the subjects treated with the SCCD demonstrate, on average, a 30% greater reduction in pain on the VAS as compared to the control subjects.

SECONDARY OUTCOMES:
Quantitative Sensation | 30 days
  1) The ability of the subject to discriminate temperature and vibration on the bottom of the foot as measured by a quantitative tool.
Analgesic Use | 30 days
  4) Improvement in PDN as measured by the change in usage of prescribed regimented and breakthrough medications for analgesia
Quality of Life | 30 days
  3) Improved quality of life as measured using the SF36 QOL questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Sean D Rosenblum DPM, Lodi, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other investigators. Data sent to the data assessor will be anonymous.